CLINICAL TRIAL: NCT07127302
Title: Evaluation and Clinical Correlation of Tendons With Power Doppler, SWE, Microvascular Flow (MV-Flow) Imaging and B-Mode Ultrasonography in Patients With Lateral Epicondylitis
Brief Title: Correlation of Ultrasonographic Findings With Clinical Parameters in Patients With Lateral Epicondylitis
Status: Recruiting | Type: Observational
Sponsor: Ahmet Yesildag (Other)
Responsible Party: Sponsor-Investigator, Ahmet Yesildag, prof. dr., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Other Study IDs: 19-2025/10
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lateral Epicondylitis; Elastography; Ultrasonographic Diagnosis; Tennis Elbow
Keywords: Lateral epicondylitis; Ultrasonographic diagnosis; Doppler Ultrasound
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Medical imaging, Patient data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation and Clinical Correlation of Tendons Using Power Doppler, SWE, Microvascular Flow (MV-Flow) Imaging and B-Mode Ultrasonography in Patients with Lateral Epicondylitis.

DETAILED DESCRIPTION:
The aim of the study was to perform tendon evaluation using different ultrasonography methods in patients with a diagnosis or prediagnosis of lateral epicondylitis and to determine the correlation between clinical findings and ultrasonographic findings. Hemodynamic and elastic properties of pathologic tendons will be examined using Power Doppler, Shear Wave Elastography (SWE), Microvascular Flow (MV-Flow) and B-Mode Ultrasonography methods.

In addition, clinical scoring of the cases will be compared with positive wrist extension tests agonist resistance (Cozen test) duration of pain in the lateral epicondyle region (weeks), VAS pain score at rest, VAS pain score during activity, VAS pain score during maximal grip, VAS pain score during maximal grip, and US findings to determine the ultrasonography technique with the highest clinical correlation.

In addition, the differences between pathologic tendons and normal tendons will be evaluated to determine the Doppler US findings with the highest diagnostic performance.

ELIGIBILITY:
Inclusion Criteria:

Lateral epicondylitis

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lateral epicondylitis or suspected lateral epicondylitis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
The relationship between clinical scores and ultrasound findings in patients with lateral epicondylitis. | 3-5 months
  Correlation or logistic statistical analyses will be applied to reveal the relationship between ultrasound methods and clinical scores.

SECONDARY OUTCOMES:
Comparison of ultrasound findings in pathological tendons and normal tendons and demonstration of the diagnostic performance of ultrasound methods | 3-5 Month
  Ultrasound measurements of normal and patological tendons will be compared by statistical methods such as indipendent T-test or Mann Whitney U.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Yeşildağ, Prof.Dr., Study Director — Karamanoğlu Mehmetbey Universty
Locations (1):
- Karamanoglu Mehmetbey Universty, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Juul-Kristensen B, Lund H, Hansen K, Christensen H, Danneskiold-Samsoe B, Bliddal H. Poorer elbow proprioception in patients with lateral epicondylitis than in healthy controls: a cross-sectional study. J Shoulder Elbow Surg. 2008 Jan-Feb;17(1 Suppl):72S-81S. doi: 10.1016/j.jse.2007.07.003. Epub 2007 Nov 26. PMID 18036844
- [Background] Zhou J, Yang DB, Wang J, Li HZ, Wang YC. Role of shear wave elastography in the evaluation of the treatment and prognosis of supraspinatus tendinitis. World J Clin Cases. 2020 Jul 26;8(14):2977-2987. doi: 10.12998/wjcc.v8.i14.2977. PMID 32775379
- [Background] Unal OF, BayramoGlu Z, AdaletlI I. Evaluation of Periarticular Soft Tissues in Patients With Juvenile Idiopathic Arthritis by Superb Microvascular Imaging and Shear Wave Elastography. Arch Rheumatol. 2020 Feb 7;35(2):264-273. doi: 10.46497/ArchRheumatol.2020.7640. eCollection 2020 Jun. PMID 32851377
- [Background] Gitto S, Messina C, Chianca V, Tuscano B, Lazzara A, Corazza A, Pedone L, Albano D, Sconfienza LM. Superb microvascular imaging (SMI) in the evaluation of musculoskeletal disorders: a systematic review. Radiol Med. 2020 May;125(5):481-490. doi: 10.1007/s11547-020-01141-x. Epub 2020 Feb 4. PMID 32020529
- [Background] Praet SFE, Ong JH, Purdam C, Welvaert M, Lovell G, Dixon L, Gaida JE, Anglim J, Manzanero S, Vlahovich N, Hughes D, Waddington G. Microvascular volume in symptomatic Achilles tendons is associated with VISA-A score. J Sci Med Sport. 2018 Dec;21(12):1185-1191. doi: 10.1016/j.jsams.2018.05.013. Epub 2018 May 15. PMID 29789266
- [Background] Arslan S, Karahan AY, Oncu F, Bakdik S, Durmaz MS, Tolu I. Diagnostic Performance of Superb Microvascular Imaging and Other Sonographic Modalities in the Assessment of Lateral Epicondylosis. J Ultrasound Med. 2018 Mar;37(3):585-593. doi: 10.1002/jum.14369. Epub 2017 Aug 29. PMID 28850740